CLINICAL TRIAL: NCT03080285
Title: Efficacy of Over-glasses Patch Treatment for Amblyopia in Children :OPTA Study, A Prospective Randomized Clinical Trial
Brief Title: Efficacy of Over-glasses Patch Treatment for Amblyopia in Children : OPTA Study
Acronym: OPTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Heeyoung Choi, Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1404-021-017
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional patch (Active Comparator): The patients were prescribed 2 hours of patching per day for the sound eye and the spectacles were to be worn full-time.
  Conventional patch is occlusion treatment sticker (Opticlude Eye Patch, 3M, Maplewood, MN, USA) with an adhesive material attached to the skin and serves to cover the eyes.
  Interventions: Device: Conventional patch
- over-glasses patch (Experimental): the patients were prescribed 2 hours of patching per day for the sound eye and the spectacles were to be worn full-time.
  Over-glasses patch (Tomato Eye Patch, Tomato Inc., Busan, South Korea) is made of fabric and covers the glasses, hence serves to cover the eyes.
  Interventions: Device: over-glasses patch

INTERVENTIONS:
Device: over-glasses patch — Over-glasses patch (Tomato Eye Patch, Tomato Inc., Busan, South Korea) is applied to the patients. They were prescribed 2 hours of patching per day for the sound eye.
  Arms: over-glasses patch
Device: Conventional patch — Conventional patch (Opticlude Eye Patch, 3M, Maplewood, MN, USA) is applied to the patients. They were prescribed 2 hours of patching per day for the sound eye.
  Arms: Conventional patch

SUMMARY:
This is a study to investigate efficacy of over-glasses patch treatment for amblyopic children using visual function improvement and Amblyopia Treatment Index (ATI) changes.

DETAILED DESCRIPTION:
In a randomized multi-center controlled clinical trial, children younger than 7 years with moderate amblyopia (visual acuity in the range of 20/40 to 20/100) would be included to receive treatment with either a conventional patch or an over-glasses patch. The patients will be prescribed 2 hours of patching per day for the sound eye. Best-corrected visual acuity (BCVA) and stereopsis will be investigated and ATI questionnaires be collected from parents at 5 weeks and 17 weeks after the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. moderate amblyopia (logMAR visual acuity in the amblyopic eye 0.3 to 0.7 inclusive)
2. logMAR visual acuity in the sound eye of 0.1 or better
3. intereye acuity difference of larger or equal to 0.3 of logMAR visual acuity
4. the presence of or a history of an amblyogenic factor meeting study-specified criteria for strabismus and/or anisometropia.

Exclusion Criteria:

1. presence of an ocular cause for low vision
2. myopia greater than -6.0 diopters (D) spherical equivalent in either eye
3. prior intraocular or refractive surgery
4. treatment for amblyopia (other than spectacle correction) within the 6 months prior to the enrollment
5. Down syndrome

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity (logMAR) | 17 weeks
  changes in best- corrected visual acuity between before treatment and after 17 weeks.
  Visual acuity is assessed using the Snellen chart. logMAR visual acuity ranges 0.0 to 3.0. logMAR visual acuity of 0.0 corresponds to 20/20. Lower scores represents better functioning.

SECONDARY OUTCOMES:
amblyopia treatment index | 17 weeks
  A modified version of ATI was provided to the parent(s) of all the enrolled minor patients as part of their follow-up visit with their child. The test consisted of 20 items, translated to Korean by one English language specialist and three ophthalmologists. The score from each question contributed to a sub-scale of the adverse effect (question numbers 2, 3, 4, 7, 8, 9, 13, and 16), compliance (question numbers 1, 5, 6a, 10 and 12), and social stigma (question numbers 11, 14 and 18). The questionnaires were scored on a 5-point Likert scale system, and the parent-provided questionnaire used a strength of agreement scale with responses of "strongly agree" (5), "agree" (4), "neither agree nor disagree" (3), "disagree" (2), "strongly disagree" (1), and "not applicable." In the test, the majority of items were negative statements, and therefore, a higher score indicated a higher negative impact or a higher burden. Reverse scoring was applied to the few items that were positive statements.
the best corrected visual acuity | 17 weeks
  best corrected visual acuity (logMAR) at 17 weeks Visual acuity is assessed using the Snellen chart. logMAR visual acuity ranges 0.0 to 3.0. logMAR visual acuity of 0.0 corresponds to 20/20. Lower scores represents better functioning.
change of binocularity | 17 weeks
  A binocularity index was determined with the use of the Worth 4 Dot test at near and the Titmus stereo test with a scale ranging from 0 to 4 with the following characteristics: 0, indicating complete suppression; 1, a moderate central suppression scotoma with peripheral fusion at near only indicated by fusion on the Worth 4 Dot test at near; 2, a small suppression scotoma and peripheral fusion indicated by fusion of the Titmus stereo fly; 3, moderate stereoacuity (100-400 arc seconds) on the stereo test animals (1 to 3 animals) and/or on the stereo test circles (1 to 5 circles); and 4, good stereoacuity (<80 arc seconds ) on the stereo test circles (6 to 9 circles).

CONTACTS AND LOCATIONS:
Overall Officials: Hee young Choi, MD, PhD, Study Chair — Pusan National University hospotal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scheiman MM, Hertle RW, Beck RW, Edwards AR, Birch E, Cotter SA, Crouch ER Jr, Cruz OA, Davitt BV, Donahue S, Holmes JM, Lyon DW, Repka MX, Sala NA, Silbert DI, Suh DW, Tamkins SM; Pediatric Eye Disease Investigator Group. Randomized trial of treatment of amblyopia in children aged 7 to 17 years. Arch Ophthalmol. 2005 Apr;123(4):437-47. doi: 10.1001/archopht.123.4.437. PMID 15824215
- [Result] Flynn JT, Schiffman J, Feuer W, Corona A. The therapy of amblyopia: an analysis of the results of amblyopia therapy utilizing the pooled data of published studies. Trans Am Ophthalmol Soc. 1998;96:431-50; discussion 450-3. PMID 10360300
- [Result] Wallace MP, Stewart CE, Moseley MJ, Stephens DA, Fielder AR; Monitored Occlusion Treatment Amblyopia Study (MOTAS) Cooperatives; Randomized Occlusion Treatment Amblyopia Study (ROTAS) Cooperatives. Compliance with occlusion therapy for childhood amblyopia. Invest Ophthalmol Vis Sci. 2013 Sep 17;54(9):6158-66. doi: 10.1167/iovs.13-11861. PMID 23882695